CLINICAL TRIAL: NCT03057626
Title: LEAHRN (Late Effects After High-Risk Neuroblastoma) Study
Brief Title: Late Effects After Treatment in Patients With Previously Diagnosed High-Risk Neuroblastoma
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ALTE15N2; NCI-2017-00170 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ALTE15N2 (Other: Children's Oncology Group); COG-ALTE15N2 (Other: DCP); ALTE15N2 (Other: CTEP); UG1CA189955 (NIH)
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Neuroblastoma; Stage 2A Neuroblastoma; Stage 2B Neuroblastoma; Stage 3 Neuroblastoma; Stage 4 Neuroblastoma; Stage 4S Neuroblastoma
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (specimen collection): Patients undergo collection of blood and urine samples on day 1. Patients also undergo clinical assessments, laboratory, radiographic, and other ancillary studies on day 1.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Undergo collection of blood and urine
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies

SUMMARY:
This research trial studies late effects after treatment in patients with previously diagnosed high-risk neuroblastoma. Studying late effects after treatment may help to decide which treatments for high-risk neuroblastoma are better tolerated with less side effects over time.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the prevalence of organ dysfunction, subsequent malignant neoplasm (SMN), growth impairment, abnormal pubertal development, and neurobehavioral dysfunction in a large cohort of representative 5-year survivors of high-risk neuroblastoma treated with modern therapy.

II. To identify the demographic, clinical and treatment-related risk factors associated with increased risk of organ dysfunction, SMN, growth impairment, abnormal pubertal development and neurobehavioral dysfunction in long-term survivors of high-risk neuroblastoma.

III. To explore the impact of new biologic therapies and diagnostics including immunotherapy, immunocytokines, isotretinoin (cis-retinoic acid) and iobenguane I-131 (131 I-MIBG) on the risk of late effects.

IV. To determine the impact of impaired organ function, physical growth, pubertal development, and neurobehavioral function on health-related quality of life (HRQOL) in long-term survivors of high-risk neuroblastoma.

SECONDARY OBJECTIVES:

I. To establish a cohort of high-risk neuroblastoma survivors, with stored peripheral blood samples, who were treated with multi-modal therapies since the year 2000 as a resource for future investigation.

OUTLINE:

Patients undergo collection of blood and urine samples on day 1. Patients also undergo clinical assessments, laboratory, radiographic, and other ancillary studies on day 1.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been enrolled on COG neuroblastoma biology study ANBL00B1
* Patient must have been diagnosed with high-risk neuroblastoma per ANBL00B1 definition
* Patient must have been diagnosed on or after January 1, 2000
* At least 5 years must have elapsed since diagnosis
* Patients must have been treated for high-risk neuroblastoma

  * Note: patients may have had any therapy for high-risk neuroblastoma, including second line or non-established therapies (for example in the setting of less than optimal initial response or concerns for high risk of relapse); patients may have received therapy for refractory or relapsed neuroblastoma, or treatment for an SMN; however all cytotoxic anti-neuroblastoma therapy should have been administered >= 2 years of the enrollment date; SMN therapy may be completed or ongoing at the time of enrollment

Exclusion Criteria:

* Patients must not be currently receiving active anti-neuroblastoma cytotoxic chemotherapy
* Patients must not have received anti-neuroblastoma cytotoxic chemotherapy within the last two years

  * Note: cytotoxic therapies include (but are not limited to) chemotherapy (platinum agents, alkylators, anthracyclines, topoisomerases, vinca alkaloids, other cytotoxic chemotherapy), any kind of transplant, MIBG therapy, and/or radiation therapy
  * Non-cytotoxic (biologic/targeted/differentiating/other) therapies are permitted at the time of enrollment; for example, patients receiving oral differentiating agents, antiangiogenic therapy, immune modulators, holistic therapies, difluoromethylornithine (DMFO), other minimal residual disease (MRD) therapies/relapse-prevention therapies are eligible
* Patients with current active neuroblastoma relapse are ineligible

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients enrolled on Children's Oncology Group (COG) study ANBL00B1 diagnosed with high-risk neuroblastoma
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of specific late effects | Up to 3 years
  Late effects of interest are organ dysfunction, subsequent malignant neoplasms (SMN), growth impairment, abnormal pubertal development, and neurobehavioral dysfunction. Prevalence will be calculated as the number of patients with late effects divided by the number with known status of that endpoint.
Risk factors of late effects | Up to 3 years
  Risk factors of interest include sex, race, ethnicity, current age, length of follow up, MYCN status, stage, primary site, age at diagnosis, total anthracycline dose (doxorubicin equivalents), cyclophosphamide dose equivalent categories, total platinum exposure (dose), topotecan exposure (yes [Y]/no [N]), cis-retinoic acid exposure (Y/N), GD-2/cytokine exposure (Y/N), radiation (Y/N), abdominal RT (Y/N), radiation to metastatic sites (Y/N), number of transplants, number of meta-iodobenzylguanidine (MIBG) scans, and therapeutic MIBG (Y/N). Will be reported as the number of patients with the risk factor divided by the number with known status of that risk factor for categorical variables and descriptively (mean, standard deviation) for continuous variables.
Pediatric Quality of Life (PedsQL) score | Up to 3 years
  PedsQL score will be reported descriptively (mean, standard deviation). The proportion of patients with impaired physical growth, delayed pubertal development, chronic disease, impaired executive functioning, and impaired social functioning will also be reported.

SECONDARY OUTCOMES:
Collection and storage of blood samples | Up to 3 years
  Proportion of survivors and their families that consent for future utilization of their banked sample for future research will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Tara O Henderson, Principal Investigator — Children's Oncology Group
Locations (98):
- United States (84):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Australia (2):
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - Perth Children's Hospital, Perth, Western Australia
- Canada (11):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec
- Starship Children's Hospital, Grafton, Auckland, New Zealand